CLINICAL TRIAL: NCT01392755
Title: A Study to Evaluate the Effects of Two Different Meal Types, Omeprazole and Ranitidine on Danoprevir Pharmacokinetics When Coadministered With Ritonavir in Healthy Subjects
Brief Title: A Study to Evaluate The Effects of Two Different Meal Types, Omeprazole And Ranitidine On Danoprevir Pharmacokinetics When Coadministered With Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25291
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Omeprazole; Ranitidine; Ritonavir

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: danoprevir; Drug: ritonavir
- 2 (Experimental)
  Interventions: Drug: danoprevir; Drug: omeprazole; Drug: ranitidine; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — oral doses of danoprevir
Drug: omeprazole — oral doses of omeprazole
  Arms: 2
Drug: ranitidine — oral dose of ranitidine
  Arms: 2
Drug: ritonavir — oral doses of ritonavir

SUMMARY:
This randomized, open-label study will evaluate the effect of food, and the effect of omeprazole and ranitidine on danoprevir co-administered with ritonavir. Volunteers will be assigned to one of two treatment groups. Volunteers in both groups will receive oral doses of danoprevir and ritonavir. In addition, volunteers in group 2 will receive oral doses of omeprazole and ranitidine. The anticipated time of the study is approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, aged 18 to 45 years, inclusive
* Weight >/= 50.0 kg
* Body Mass Index (BMI) 18.0 to 32.0 kg/m2, inclusive

Exclusion Criteria:

* Presence of any active or chronic disease
* Abnormal blood pressure
* Abnormal resting heart rate
* Abnormal ECG values
* History of any clinically significant cardiovascular or cerebrovascular disease
* Current smokers or subjects that have discontinued smoking < 6 months prior to first dose of study drug
* Positive for hepatitis B, hepatitis C or HIV
* Positive test for drugs of abuse or alcohol
* Positive result for H. pylori
* Regular use of antacids, H-2 blockers, proton pump inhibitors, or any investigational drug within 30 days of first dose of study medication
* History of clinically significant gastrointestinal disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Effect of omeprazole on the area under the plasma concentration time curve of danoprevir when co-administered with ritonavir | 1 day
Effect of ranitidine on the area under the plasma concentration time curve of danoprevir when co-administered with ritonavir | 1 day
Food effect on area under the plasma concentration time curve of danoprevir when co-administered with ritonavir | 1 day

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | Approximately 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States